CLINICAL TRIAL: NCT06743750
Title: Comparison Between Nasopharynx and Orobuccal/Nasal Swabs or Saliva for Detection of Respiratory Viruses (ORASAMP)
Brief Title: Comparison Between Different Sampling Sites for Detection of Respiratory Viruses
Acronym: ORASAMP
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 5888
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Tract Infection Viral
Keywords: Viral respiratory tract infection; Diagnostic test performance; Molecular diagnostic; Influenza; RSV; Rhinovirus
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Orobuccal and nasal swab as well as saliva will be retained until the end of the study. For participants agreeing to further analyses of the samples with an additional consent, samples will be stored up to a maximum of 10 years after the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study sample: There is only one group in this study
  Interventions: Diagnostic Test: RT-PCR in different respiratory tract samples

INTERVENTIONS:
Diagnostic Test: RT-PCR in different respiratory tract samples — RT-PCR on saliva, orrobuccal swab and nasal swab will be performed. Nasopharyngeal swab will be performed independently of the study as standard of care.

SUMMARY:
The goal of this observational study is to validate the use of less invasive samples (saliva, orobuccal or nasal swabs) than nasopharyngeal swab for testing common and clinically relevant respiratory viruses in children and adults presenting to an emergency departements with symptoms compatible with respiratory tract infection. The main question it aims to answer is:

- Is the precision of reverse transcription polymerase chain reaction (RT-PCR) for Influenzavirus A or B, respiratory syncytial virus (RSV), and Rhinovirus, on saliva, orobuccal swabs and nasal swabs comparable to the gold standard nasopharyngeal swab in a pediatric and adult population presenting with symptoms compatible with respiratory tract infection.

Among participants the following samples will be collected (nasopharyngeal swab is standard of care and not part of the study samples):

* Saliva
* Orobuccal swab
* Nasal swab

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at the emergency departments or hospitalized at Inselspital Bern university hospital with any symptom compatible with an acute respiratory tract infection in whom a nasopharyngeal swab to test for respiratory viruses is performed (standard of care)
* Written informed consent from the trial subject has been obtained; for patients aged 0-13 years, or not able to provide informed consent, consent obtained from the legal representative; for patients between 14-18 years, written informed consent obtained from the respective patient as well as the legal representative.

Exclusion Criteria:

* Patients unable to provide a saliva (e.g. patients with reduced level of consciousness). Children too young to be instructed to provide saliva are not excluded, but saliva won't be collected.
* Patients with swallowing disturbances
* Patient's lack of accountability and inability to appreciate the nature, meaning and consequences of the study and to formulate his/her own wishes correspondingly AND legal representative not available.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children or adults presenting at the emergency departments or hospitalized at the University Hospital of Bern with any symptom compatible with an acute respiratory tract infection in whom a nasopharyngeal swab to test for respiratory viruses is performed (standard of care).
  Consecutive participant recruitment will be performed at the children and adult emergency departments during working hours of the study nurse.
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Sensitivity of RT-PCR for Influenzavirus A or B, RSV and Rhinovirus, on orobuccal or nasal swab and saliva compared to nasopharyngeal swab. | At baseline
Specificity of RT-PCR for Influenzavirus A or B, RSV and Rhinovirus, on orobuccal or nasal swab and saliva compared to nasopharyngeal swab. | At baseline

SECONDARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve for the detection of Influenza A/B, RSV and Rhinovirus in each study sample (orobuccal or nasal swab and saliva). | At baseline
Positive agreement between viral copy number of RT-PCR for Influenzavirus A or B, RSV, and Rhinovirus, Parainfluenzavirus, Adenovirus, human Metapneumovirus in saliva, orobuccal swabs and nasal swabs compared to nasopharyngeal swabs. | At baseline
Negative agreement between viral copy number of RT-PCR for Influenzavirus A or B, RSV, and Rhinovirus, Parainfluenzavirus, Adenovirus, human Metapneumovirus in saliva, orobuccal swabs and nasal swabs compared to nasopharyngeal swabs. | At baseline
Prevalence of respiratory viruses in orobuccal, nasal or nasopharyngeal swabs and saliva. | At baseline
Sensitivity of RT-PCR for Parainfluenzavirus, Adenovirus and human Metapneumovirus in orobuccal, nasal and saliva samples. | At baseline
Specificity of RT-PCR for Parainfluenzavirus, Adenovirus and human Metapneumovirus in orobuccal, nasal and saliva samples. | At baseline
Incremental yield of virus detection in orobuccal, nasal and saliva as compared to nasopharyngeal samples. | At baseline
Co-prevalence of respiratory viruses in orobuccal, nasal or nasopharyngeal swabs and saliva. | At baseline
Association between predefined symptoms and probability for positive RT-PCR of specific viruses using different (nasopharyngeal, orobuccal, nasal, saliva) samples. | At baseline
Comparative cycling time values at the different sampling locations | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Jent, MD, Principal Investigator — University Hospital of Bern, University of Bern
Locations (1):
- Inselspital, University Hospital of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No